CLINICAL TRIAL: NCT06735651
Title: Wild Blueberries for Gut, Brain, and Cardiometabolic Health in Female Adults With Prediabetes.
Brief Title: Wild Blueberries for Gut, Brain, and Cardiometabolic Health in Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Principal Investigator, Rafaela G. Feresin, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H24123
Record Dates: First submitted 2024-11-05; First posted 2024-12-16 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Female; Adult; Endothelial Function (Reactive Hyperemia); Arterial Stiffness; Cognition; Oxidative Stress; Gut Microbiota; Overweight; Inflammation; Microvascular Function; Body Composition
Keywords: Blueberries; Prediabetes; Insulin Resistance; Functional foods; Dietary intervention; Endothelial function; Vascular function; Cardiovascular health; Metabolic health; Gut microbiota; Cognitive function; Type II diabetes; Microvascular Function; Wild Blueberries
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance; Hyperemia; Overweight; Inflammation; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wild Blueberry (Experimental): 22 g of freeze-dried wild blueberry freeze-dried powder per day
  Interventions: Dietary Supplement: Wild Blueberry
- Placebo (Placebo Comparator): 22 g of freeze-dried macronutrient-matched placebo powder per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wild Blueberry — Daily consumption of 22 g of freeze-dried wild blueberry freeze-dried powder for 6 weeks
  Arms: Wild Blueberry
Dietary Supplement: Placebo — Daily consumption of 22 g of freeze-dried macronutrient-matched placebo powder for 6 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of using a freeze-dried wild blueberry powder on cardiometabolic health, cognitive function, and gut microbiota composition in adult women with prediabetes.

DETAILED DESCRIPTION:
In the U.S., 35.3 million adults have type 2 diabetes mellitus (T2DM) and 96 million have prediabetes. Eight out of 10 people with T2DM die from cardiovascular disease. People with T2DM also have a 50% higher risk of developing dementia compared to healthy counterparts. Further, studies show that gut microbes play a major role in the development of T2DM. Prevention and treatment of T2DM focus on lifestyle changes including dietary modifications such as increased consumption of deep-colored fruits like berries. Blueberries are rich in fiber and phytochemicals and have several health benefits. We and others have shown that blueberry intake improves heart health in healthy men, hypertensive postmenopausal women, and men and women with metabolic syndrome. Yet, a comprehensive study in women with prediabetes that measures changes in cognitive performance and the underlying heart and gut health has not been conducted to date. Thus, the overall objective of this study is to investigate and bring forth evidence that wild blueberries improve gut, cardiometabolic, and cognitive function in women with prediabetes.

Therefore, this pilot six-week randomized, placebo-controlled parallel-arm clinical trial aims to investigate whether daily consumption of 22 g of freeze-dried wild blueberry powder improves gut, cardiometabolic, and cognitive function in women with prediabetes. Investigators hypothesize that daily consumption of wild blueberries will improve cardiometabolic parameters, gut dysbiosis, and cognitive impairments in our study population. To test these hypotheses, the following specific aims are proposed. To investigate whether daily consumption of 22 g of freeze-dried wild blueberry powder:

* Reduces levels of fasting blood glucose (FBG), insulin, and HOMA-IR (homeostatic model assessment of insulin resistance) and improves lipid profile in women with prediabetes.
* Reduces blood pressure and improves endothelial function in women with prediabetes.
* Improves cognitive function (verbal memory and executive functions [inhibition, working memory, cognitive flexibility]) in women with prediabetes.
* Favorably modulates gut microbiota composition in women with prediabetes.
* Improves serum markers of oxidative stress and inflammation in women with prediabetes.

Additionally, whether changes in the gut microbiota are associated with changes in cardiometabolic and cognitive function outcomes and whether changes in cardiometabolic outcomes are associated with changes in cognitive function parameters will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-65 years old
* Prediabetes (fasting blood glucose 100-125 mg/dL and/or HbA1c percentage between 5.7-6.4)
* Body Mass Index between 25-30 kg/m^2

Exclusion Criteria:

* Allergies to berries
* Use of insulin, antidiabetic, antibiotics, and anti-inflammatory drugs
* Active cancer, gastrointestinal, renal, thyroid, stage 1 & 2 hypertension and other cardiovascular diseases, neurological diseases, or severe head injury
* Smoking
* Consumes greater than 2 alcoholic beverages per day
* Consumes antioxidant, probiotic, and prebiotic supplements
* Pregnant or Lactating
* Actively participating in a weight loss program
* Currently taking berry supplements or recently participated in another study taking berry supplements

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | Baseline and 6 weeks
  Measurement of fasting blood glucose
Ambulatory Blood Pressure | Baseline and 6 weeks
  Assessment of whole-day ambulatory blood pressure during daytime and nighttime periods.

SECONDARY OUTCOMES:
Fasting Insulin | Baseline and 6 weeks
Homeostasis model assessment-insulin resistance (HOMA-R) | Baseline and 6 weeks
  Calculated as fasting insulin (mU/mL) x fasting glucose (mg/dL)/405
Blood Lipid Profile | Baseline and 6 weeks
  Measurement of blood lipid profile
Gut Microbiota Composition | Baseline and 6 weeks
  Analysis of stool sample for determination of absolute levels of bacteria and relative species composition
Global Cognitive Ability | Screening
  Measured using NIH Toolbox Picture Vocabulary test and Oral Reading Recognition
Performance Validity | Baseline and 6 weeks
  Assessed using Rey 15
Verbal Memory & Recognition | Baseline and 6 weeks
  Measured using Rey Auditory Verbal Learning Test with appropriate alternate forms
Cognitive Inhibition | Baseline and 6 weeks
  Measured using Delis-Kaplan Executive Function System Color Word Interference, and NIH Toolbox Flanker Inhibitory Control and Attention
Cognitive Flexibility | Baseline and 6 weeks
  Assessed using Delis-Kaplan Executive Function System Trails and Verbal Fluency Switching
Working Memory | Baseline and 6 weeks
  Measured using Digit Span and NIH Toolbox List Sorting
Processing Speed | Baseline and 6 weeks
  Measured using NIH Toolbox Pattern Comparison and Oral Symbol Digit tests
Associative Memory | Baseline and 6 months
  Measured using NIH Toolbox Face Name Associative Memory Exam and Face Name Associative Memory Exam Delay tests
Attention | Baseline and 6 weeks
  Assessed using Wechsler Adult Intelligence Scale - IV and Rey Auditory Verbal Learning Test Trial 1.
Problem-Solving | Baseline and 6 weeks
  Assessed using NIH Toolbox Visual Reasoning Test

OTHER OUTCOMES:
Reactive Hyperemia Index | Baseline and 6 weeks
  Assessment of endothelial function in response to increased shear stress using EndoPAT2000
Pulse Wave Velocity | Baseline and 6 weeks
  Arterial Stiffness will be assessed by pulse wave velocity using SphygmCor
Percent Maximal Microvascular Blood Flow | Baseline and 6 weeks
  Micro-vessel blood flow in response to local heating stimulus will be assessed using a Laser Doppler
Circulating Markers of Inflammation and Oxidative Stress | Baseline and 6 weeks
  Measurement of concentrations of circulating markers of inflammation such as CRP and oxidative stress such as TBARS in blood plasma and serum samples.
Urinary Polyphenolic Metabolites | Baseline and 6 weeks
  24-hour urine collection samples will be assessed for polyphenol metabolites
Body Fat | Baseline and 6 weeks
  DEXA will be used to assess body fat.

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela G Feresin, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stote KS, Wilson MM, Hallenbeck D, Thomas K, Rourke JM, Sweeney MI, Gottschall-Pass KT, Gosmanov AR. Effect of Blueberry Consumption on Cardiometabolic Health Parameters in Men with Type 2 Diabetes: An 8-Week, Double-Blind, Randomized, Placebo-Controlled Trial. Curr Dev Nutr. 2020 Mar 9;4(4):nzaa030. doi: 10.1093/cdn/nzaa030. eCollection 2020 Apr. PMID 32337475
- [Background] Miller MG, Hamilton DA, Joseph JA, Shukitt-Hale B. Dietary blueberry improves cognition among older adults in a randomized, double-blind, placebo-controlled trial. Eur J Nutr. 2018 Apr;57(3):1169-1180. doi: 10.1007/s00394-017-1400-8. Epub 2017 Mar 10. PMID 28283823
- [Background] Biessels GJ, Despa F. Cognitive decline and dementia in diabetes mellitus: mechanisms and clinical implications. Nat Rev Endocrinol. 2018 Oct;14(10):591-604. doi: 10.1038/s41574-018-0048-7. PMID 30022099
- [Background] Rawshani A, Rawshani A, Franzen S, Eliasson B, Svensson AM, Miftaraj M, McGuire DK, Sattar N, Rosengren A, Gudbjornsdottir S. Mortality and Cardiovascular Disease in Type 1 and Type 2 Diabetes. N Engl J Med. 2017 Apr 13;376(15):1407-1418. doi: 10.1056/NEJMoa1608664. PMID 28402770
- [Background] Krikorian R, Skelton MR, Summer SS, Shidler MD, Sullivan PG. Blueberry Supplementation in Midlife for Dementia Risk Reduction. Nutrients. 2022 Apr 13;14(8):1619. doi: 10.3390/nu14081619. PMID 35458181
- [Background] Johnson SA, Figueroa A, Navaei N, Wong A, Kalfon R, Ormsbee LT, Feresin RG, Elam ML, Hooshmand S, Payton ME, Arjmandi BH. Daily blueberry consumption improves blood pressure and arterial stiffness in postmenopausal women with pre- and stage 1-hypertension: a randomized, double-blind, placebo-controlled clinical trial. J Acad Nutr Diet. 2015 Mar;115(3):369-377. doi: 10.1016/j.jand.2014.11.001. Epub 2015 Jan 8. PMID 25578927